CLINICAL TRIAL: NCT05375604
Title: Phase 1 Study of Macrophage Reprogramming Agent, exoASO-STAT6 (CDK-004), in Patients With Advanced Hepatocellular Carcinoma (HCC) and Patients With Liver Metastases From Either Primary Gastric Cancer or Colorectal Cancer (CRC)
Brief Title: A Study of exoASO-STAT6 (CDK-004) in Patients With Advanced Hepatocellular Carcinoma (HCC) and Patients With Liver Metastases From EIther Primary Gastric Cancer or Colorectal Cancer (CRC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Bankruptcy
Sponsor: Codiak BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDK-004-101
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC); Gastric Cancer Metastatic to Liver; Colorectal Cancer Metastatic to Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental CDK-004 (Experimental): CDK-004 administered as a single agent intravenously (IV) on Days 1 and 15 of Cycles 1 and 2, on Day 1 of every Cycle.
  Interventions: Drug: CDK-004

INTERVENTIONS:
Drug: CDK-004 — ASO-STAT6 exosome administered Intravenously
  Other Names: exoASO-STAT6

SUMMARY:
This is a first-in-human, Phase 1 open-label, multicenter, dose escalation, safety, pharmacodynamic, and PK study of exoASO-STAT6 (CDK-004) in patients with advanced Hepatocellular Carcinoma (HCC) and patients with liver metastases from either primary gastric cancer or colorectal cancer (CRC).

DETAILED DESCRIPTION:
CDK-004 as an intravenous (IV) treatment for advanced hepatocellular carcinoma (HCC), and primary gastric cancer or CRC with secondary liver metastases.

CDK-004 is an investigational therapeutic candidate consisting of cell-derived exosomes loaded with a synthetic lipid-tagged oligonucleotide.

CDK-004 is designed to allow for specific delivery of the STAT6 anti-sense oligonucleotide (ASO) to the myloid to repolarize macrophage from immune suppressive M2 to proinflammatory M1 phenotype, with a potential for meaningful single agent antitumor activity which has not been observed with other pathway inhibitors to date.

CDK-004 will be administered as a single agent intravenously (IV) at various doses.

Dose limiting toxicities (DLTs) will be assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Must have one of the following cancer types:

   1. Advanced HCC defined as Barcelona Clinic Liver Cancer (BCLC) Stage B/C not amenable to resection or locoregional therapy;
   2. Histologic or radiologic proof of liver metastasis from primary CRC which is unresectable with no evidence of extrahepatic metastasis;
   3. Histologic or radiologic proof of liver metastasis from primary gastric cancer which is unresectable with no evidence of extrahepatic metastasis.
2. Documented progression after at least 1 line of FDA approved systemic therapy for advanced HCC/gastric cancer/CRC or intolerable/refuse to chemotherapy.
3. ≥ 18 years of age at screening.
4. Measurable disease by RECIST v1.1.
5. Able to provide archival tumor tissue/fresh biopsy prior to study treatment and on-treatment tumor biopsies if considered safe and medically feasible by the Investigator.
6. ECOG performance status of 0-2.
7. Acceptable liver function
8. Acceptable renal function
9. Acceptable hematologic status
10. Cirrhosis classified as Child-Pugh Class A (applicable only to patients diagnosed with cirrhosis)..
11. Women of child-bearing potential agree to use highly effective contraceptive methods and avoid egg donation and preservation during the study treatment and for 6 months after the last dose of study drug.
12. Men of child-producing potential agree to use highly effective contraceptive methods and avoid sperm donation and preservation during the study treatment and for 6 months after the last dose of study drug.

Exclusion Criteria:

1. Treatment with any systemic or liver-directed anticancer therapy within 3 weeks of the first dose of study drug.
2. Uncontrolled partial or complete biliary obstruction.
3. Left ventricular ejection fraction (LVEF) < 50% at Screening.
4. 12-lead ECG demonstrating QT interval corrected by Fridericia's formula (QTcF) > 480 ms or history of long QTc syndrome.
5. Ongoing, clinically significant AEs due to prior anticancer therapies.
6. Patients with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present or in the opinion of the Investigator will not affect patient outcome.
7. Known clinically active brain metastases or known carcinomatous meningitis/leptomeningeal disease.
8. Known clinically significant infection.
9. Known clinically significant cardiac disease, including unstable angina or has had a procedure to address the underlying cause and has experienced angina within 4 weeks prior to Cycle 1 Day 1, acute myocardial infarction within 6 months from Day 1 of study drug administration, or New York Heart Association Class III or IV congestive heart failure.
10. Known history of human immunodeficiency virus (HIV).
11. If history of concurrent Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection, meets the following criteria: patients with detectable hepatitis B surface antigen (HbsAg) or detectable HBV DNA should be managed per local treatment guidelines. Controlled (treated) hepatitis B patients will be allowed if they started treatment at the time of consent and treatment is continued during study participation; patients with hepatitis C and detectable RNA are eligible if antiviral therapy has been completed prior to first administration of study drug. Testing does not need to be conducted at Screening if results from testing within the past 12 months are available.
12. History of liver transplant.
13. History of immunodeficiency or is receiving chronic systemic steroid therapy
14. Poorly controlled diabetes mellitus.
15. Active or previously documented autoimmune or inflammatory diseases
16. Is currently participating in a study of an investigational therapy or device or has participated and received an investigation therapy or device within 3 weeks of administration of CDK-004.
17. Has another physical or mental health disorder that might cause difficulty in obtaining informed consent and/or participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of CDK-004. | Up to 2 years
  Incidence of treatment-emergent adverse events as assessed by CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No